CLINICAL TRIAL: NCT05805969
Title: Efficacy of Accommodating Variable-Resistance Training on Muscle Architecture, Strength, and Functional Performance in Patients With Juvenile Idiopathic Arthritis: A Randomized Controlled Trial
Brief Title: Accommodating Variable-Resistance Training in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0036
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Intervention Model Description: A prospective, dual-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accommodating variable-resistance training (Experimental): Participants in this group received the Accommodating variable-resistance program in addition to the standard physical therapy.
  Interventions: Other: Accommodating variable-resistance training
- Standard Physical Therapy (Active Comparator): Participants in this group received the standard exercise program.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Accommodating variable-resistance training — The training was conducted twice weekly for six successive weeks under the close supervision of a licensed pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  The training protocol included maximum voluntary concentric knee flexor/extensor actions. Three sets of five to 10 repetitions of maximum-effort concentric action at angular speeds of 240, 180, and 120 degrees/second.
  The training started with a 10-minute warm-up exercise and ended up with a 5-minute cool-down exercise.
  Arms: Accommodating variable-resistance training
Other: Standard physical therapy — The program encompassed the standard exercises for patients with juvenile idiopathic arthritis (aerobic, weight-bearing, proprioceptive, flexibility, and strengthening exercises). The training was conducted for 45 minutes, two times a week for six successive weeks.
  Arms: Standard Physical Therapy

SUMMARY:
This study was designed to investigate the effect of six weeks of accommodating variable-resistance training on muscle architecture, muscle strength, and functional performance in patients with juvenile idiopathic arthritis. Fifty-eight children with juvenile idiopathic arthritis were randomly allocated to the experimental group (n = 29, received the accommodating variable-resistance training) or the Control group (n = 29, received usual physical rehabilitation alone). Both groups were assessed for muscle architecture, muscle strength, and functional performance before and after treatment.

DETAILED DESCRIPTION:
Fifty-eight patients with juvenile idiopathic arthritis participated in the study. They were recruited from King Khalid Hospital and two other referral hospitals, in Riyadh, Saudi Arabia. They were between 12 and 18 years old, had poly-articular onset and bilateral knee involvement, were on stable doses of medications, and were not engaging in regular exercise regimens. Patients were excluded if they had fixed deformities, a history of joint surgery, or whose radiological investigations revealed erosive changes of bone, ankylosing, or fractures.

Outcome measures

1. Muscle architecture: the fascicle length, pennation angle, and thickness of the vastus lateralis muscle were assessed using a standard high-resolution ultrasound imaging system.
2. Muscle strength: The peak concentric torque of the right and left knee extensors was measured through an isokinetic dynamometer.
3. Functional capacity: Three tests were used; the 6-minute walk test, the timed up and down stairs test, and the 4x10 meter Shuttle Run test.

The experimental group received a 6-week accommodating variable-resistance training, two times a week for six consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The training protocol included maximum voluntary concentric knee flexor/extensor actions through a motion range between 10 and 90 degrees. Three sets of five to 10 repetitions at angular speeds of 240, 180, and 120 degrees/second were performed. The training started with a warm-up for 10 minutes and ended with a cool-down for 5 minutes.

The control group received the standard exercise program, 45 minutes per session, two times a week for six consecutive weeks. The program consisted of flexibility exercise, strength training, weight-bearing, proprioceptive training, and free treadmill walking or cycle ergometry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of JIA
* Polyarticular onset of JIA with bilateral involvement of the knee joint
* Age between 12 and 18 years
* Stable conditions (i.e., receive stable doses of medications in the past three months)
* Not participating in a regular exercise program in the past six months

Exclusion Criteria:

* Fixed deformities
* History of joint surgery
* Ankylosing or fractures
* Bone destruction (erosive changes of the knee joint)
* Cardiopulmonary comorbidities
* Recommendation against engaging in potentially explosive physical activities by the attending Rheumatologist.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Fascicle length | 2 months
  The linear distance (mm) between the insertion into the deep and superficial aponeurosis.
Pennation angle | 2 months
  The angle (in degrees) between the fascicle and the deep aponeurosis.
Muscle thickness | 2 months
  The perpendicular distance (mm) between the deep and superficial aponeurosis.
Muscle strength | 2 months
  Indicated by the peak concentric torque of the knee extensors (Nm). It was measured using an Isokinetic Dynamometer.

SECONDARY OUTCOMES:
Six-minute walk test | 2 months
  This test identified the maximum distance (m) that each patient was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage.
Timed up and down stairs test | 2 months
  This test measured the time (seconds) that each patient took to climb up and down a 14-step stair flight (each 20 cm in height). Better performance is indicated by a shorter time.
4x10 meter Shuttle Run test | 2 months
  This test measured the time (seconds) that each patient took to run forth and back a 10-meter track. Better performance is indicated by a shorter time.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No